CLINICAL TRIAL: NCT04754061
Title: PSilocybin for psYCHological and Existential Distress in PALliative Care (PSYCHED-PAL): A Multi-site, Open-label, Single Arm Phase I/II Proof-of-concept, Dose-finding, and Feasibility Clinical Trial
Brief Title: PSilocybin for psYCHological and Existential Distress in PALliative Care (PSYCHED-PAL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Bruyère Health Research Institute. (Other); The Ottawa Hospital (Other); St. Joseph's Healthcare Hamilton (Other); CHU de Quebec-Universite Laval (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Jewish General Hospital (Other); William Osler Health System (Other); Queen's University (Other)
Responsible Party: Principal Investigator, James Downar, Head, Division of Palliative Care, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7745629246
Record Dates: First submitted 2020-11-11; First posted 2021-02-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Depression, Anxiety; Distress, Emotional
Keywords: existential distress; psychological distress; psilocybin; microdosing
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: The study is a multi-site, open-label, single-arm phase 1/2 proof-of-concept dose-finding, feasibility and preliminary efficacy clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psilocybin Microdosing (Experimental): Participants will receive a 4-week psilocybin microdosing intervention (1-3mg/day, Monday-Friday for up to 4 weeks; start at 1mg with opportunity to increase dose each week)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Phase 1 (week 1): all enrolled participants will take a single 1mg oral dose of psilocybin once per day on Monday and Thursday. If no adverse events are reported at any point during the week (Mon-Fri), the participant will continue to Phase 2 for week 2.
  Phase 2: The participant will take a single 1mg oral dose of psilocybin once per day for 5 consecutive days (Monday to Friday). If no adverse events are reported at any point during the week (Mon-Fri), the participant will continue to Phase 3 for week 3.
  Phase 3: The participant will take two 1mg oral doses (2mg total) of psilocybin once per day for 5 consecutive days (Monday to Friday). If no adverse events are reported at any point during the week (Mon-Fri), the participant will continue to Phase 4 for week 4.
  Phase 4 (maximum allowable dose): The participant will take three 1mg oral doses (3mg total) of psilocybin once per day for 5 consecutive days (Monday to Friday).

SUMMARY:
The goal of this multi-centre phase I/II open-label, single-arm study is to determine the safety, feasibility, therapeutic dose, and preliminary efficacy of psilocybin microdosing to treat psychological distress among patients with advanced illness. Forty patients will receive psilocybin drug product (1-3mg per day, Mon-Fri) for 4 weeks to be administered via oral capsules by the participant. Feasibility (recruitment rate, rate of intervention and follow-up completion), safety (rate of adverse events), dosing, and preliminary efficacy (depression, anxiety, overall well-being, and global impression of change) will be measured.

DETAILED DESCRIPTION:
Patients with advanced illness report feeling a sense of hopelessness, loss of autonomy and relationships, and a lack of purpose in life. These feelings of psychological suffering have been described as "existential distress" and are associated with poor outcomes, including decreased medication adherence and quality of life, increased desire for hastened death and rates of suicide, and has been identified as a primary reason why individuals pursue medical assistance in dying (MAiD).

Current treatments for psychological and existential suffering have low efficacy and are challenging to use in a palliative context. Pharmacological approaches for treating psychological suffering may reduce symptoms of depression and anxiety, but evidence to support their efficacy in palliative care (PC) is underwhelming. Antidepressant and anxiolytic medications also take time to work and can cause serious side effects such as falls and confusion, which can be substantial deterrents for patients. Similarly, results from randomized controlled trials (RCTs) and meta-analyses have demonstrated psychotherapeutic interventions show limited benefit in a PC population. Further, psychotherapy can be time consuming and slow to work, which is not ideal for patients with limited life expectancy. Given the burden of psychological and existential distress among patients followed by PC providers, there is a need to develop scalable, brief, and rapidly effective therapeutic approaches to reduce this distress.

Psychedelic medications offer an innovative, safe, complementary approach to address psychological and existential suffering in patients receiving PC. Studies from the 1950's showed serotonergic hallucinogens ("psychedelics") improved depression and anxiety symptoms in cancer patients. However, legislative changes restricted the use of these medications in clinical care and research. Interest in psychedelic medications has been rekindled by two recently published RCTs that studied the use of psilocybin (a mushroom-derived 5HT2A agonist) during a single psychotherapeutic session in cancer patients with anxiety and/or depression. These trials demonstrated rapid, clinically meaningful, and long-lasting reductions in depressed mood and/or anxiety symptoms and improvements in quality of life and death acceptance. There is also evidence suggesting psilocybin microdosing - taking sub-hallucinogenic doses continuously over longer time periods, rather than a one-time hallucinogenic dose - can improve mood and anxiety. The effects of microdosing, however, have not been rigorously evaluated, particularly in patients with life limiting illness.

Results from recent trials are encouraging but knowledge gaps remain. First, studies to date primarily enrolled patients with localized disease who experience different distress than that of patients with advanced disease who are near the end of life. Second, it is unclear if Canadians would find psilocybin an attractive option in the context of MAiD legalization, which provides an alternative option for patients with severe psychological suffering. Third, there is no empirical research on the therapeutic effects of psilocybin microdosing, as most studies have followed macrodosing protocols. While preliminary efficacy of macrodosing has been demonstrated, there are important barriers to administering this therapy in a PC context. Previous trials had slow recruitment rates, suggesting there may be barriers related to the acceptability of psilocybin macrodosing from the perspectives of patients and families. Macrodosing requires the patient to dedicate an entire day to participating in a guided hallucinogenic experience and remain in an acute care setting where they can be closely monitored. It also requires patients to engage in preparatory sessions with monitors and a post-therapy session. In a PC context, this time commitment may not be acceptable or feasible for patients who are nearing the end of life. Additionally, macrodosing requires at least two trained moderators to guide the patient through their psychedelic experience and facilitate the pre- and post-dosing sessions. In most PC settings, it is not feasible to have clinicians dedicate two days to a single patient, thus limiting the scalability of this intervention.

Psilocybin microdosing has the potential to overcome barriers to the feasibility and acceptability of macrodosing. By removing the requirement for trained moderators, minimizing the time commitment required of patients, eliminating the hallucinogenic effects of the therapy, and allowing patients to receive treatment either as an inpatient or in the community, microdosing may be a more acceptable option to patients and families and allow psychedelic therapy to be scalable across various PC settings. Psilocybin microdosing is a novel, complementary therapy that, while still unproven for patients near the end of life, has the potential to fundamentally change the way psychological and existential distress is responded to in PC, improving the lives of the 30% of patients who experience this suffering at the end of life.

Objective

To determine if psilocybin microdosing is a safe and feasible treatment for psychological distress among patients nearing the end of life followed by palliative care providers. All participants will receive a 4-week psilocybin microdosing intervention. The secondary objective is to examine the preliminary efficacy of psilocybin microdosing.

Sample Size

As this is a feasibility study, no formal sample size calculation was performed to determine the number of patients required to reach a level of precision on any study endpoint. Rather, the goal of this study is to provide estimates, along with their margins of error, of the recruitment rate and efficacy outcomes which will inform a subsequent two-arm randomized controlled trial. Participating sites see approximately 5,300 patients per year. It is anticipated that 30% will have psychological distress. Assuming a minimum of 1 in 6 patients are eligible and 15% of eligible patients will enroll, the goal is to enroll a sample of 20 participants in up to 1-year period.

Statistical Analysis

Analyses will adopt an intent-to-treat approach. Because the goal of this trial is to demonstrate feasibility and preliminary measures of efficacy, the main analyses will include calculation of feasibility outcomes using descriptive statistics and 95% confidence intervals (CIs), as well as effect sizes with 95% CIs for primary and secondary efficacy measures, comparing patients' 4-week follow-up assessments to baseline assessments. Participants will also be stratified based on demographic and clinical characteristics to assess trends in outcomes. Notably, there is some evidence that selective serotonin reuptake inhibitors (SSRIs) in particular may attenuate the effects of psilocybin. As such, sub-analyses will evaluate outcomes in participants taking an SSRI medication versus those who are not. A sub-group analysis by setting of care (inpatient vs outpatient/community) will also be conducted.

Analyses of safety data will include the mean and standard deviation of the peak effect observed (i.e. highest observed blood pressure, heart rate) and proportion of participants experiencing adverse mood and behaviour events. The incidence of delirium and serotonin syndrome will also be recorded.

Details of Eligibility, Intervention Protocol, and Outcome Measures are provided elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >/=18 years of age
2. Advanced illness under palliative care management, defined as having 1 to <12 months life expectancy (in the judgment of the palliative care provider)
3. Experiencing psychological distress, defined as a score of 7 or greater on the Depression, Anxiety or Well-being item of the Edmonton Symptom Assessment System
4. Ability to understand and communicate in English or French

Exclusion Criteria:

1. Current or previously diagnosed, or first-degree relative, with psychotic or bipolar disorder
2. Previously deemed eligible for MAiD with intention to proceed with MAiD regardless of study intervention effectiveness (this criteria is meant to exclude patients who would be unlikely to complete follow-up - those considering or being assessed for MAiD will still be eligible)
3. Documented or suspected delirium in the past 3 months without a clearly defined reversible cause (e.g. opioid toxicity, infection) and resolution
4. Documented moderate or severe dementia diagnosis
5. Inability to provide first-person informed consent
6. Severe or unstable physical symptoms based on the judgment of the palliative care provider
7. Palliative Performance Scale <30%
8. Cancer with known central nervous system (CNS) involvement or other CNS disease
9. Use of high-dose psychedelic substances in the past year
10. Taking lithium at any dose
11. Taking tramadol at any dose
12. Taking any monoamine oxidase inhibitor at any dose [American Hospital Formulary Service (AFHS) group 28:16.04.12 or 28:36.32, including, but not limited to, moclobemide, tranylcypromine, phenelzine, selegiline, rasagiline]
13. Taking any atypical antipsychotic (aripiprazole, asenapine, brexpiprazole, clozapine, lurasidone, olanzapine, paliperidone, quetiapine, risperidone, ziprasidone) (patients can be included if their atypical antipsychotic is either stopped, or if appropriate, substituted with haloperidol 48 hours prior to the start and for the duration of the intervention period and follow-up)
14. Inability to ingest oral capsule
15. Pregnancy or lactation

For participants taking either an SSRI or an antipsychotic medication, there are several conditions for participation: (1) the PC provider must approve their participation in the study; (2) the SSRI/anti-psychotic medication dose cannot change for the duration of the intervention trial and follow-up, and; (3) the patient must not be taking more than the maximum allowable trial dose for each SSRI.

All trial participants must agree to not take any other psychedelic substance for the duration of the clinical trial and follow-up, and to notify the investigative team of any medication changes during intervention or follow-up. Participants must also agree not to take their benzodiazepine or antipsychotic medication, if applicable, within 12 hours (6 hours pre and 6 hours post) of taking their psilocybin dose (participants will be given detailed instructions about this in their Instruction Leaflet). Participants must also agree not to drive or operate any heavy machinery on any treatment day for the duration of the 4-week intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, up to 1 year
  Number of patients enrolled divided by number of patients approached
Intervention Completion Rate | Through study completion, up to 13 months
  Number of participants who complete the intervention divided by number of participants enrolled
Follow-up Completion Rate | Through study completion, up to 18 months
  Number of participants who complete follow-up divided by number of participants enrolled
Number of Participants With Adverse Events - Change in Blood Pressure | Measured at baseline and daily (Mon-Fri) from enrolment to intervention completion (up to 4 weeks)
  Proportion of participants with systolic blood pressure of >180mmHg or an increase in 40% from baseline measurements
Number of Participants With Adverse Events - Change in Heart Rate | Measured at baseline and daily (Mon-Fri) from enrolment to intervention completion (up to 4 weeks)
  Proportion of participants with resting heart rate >100bpm or an increase in 40% from baseline
Number of Participants With Adverse Events - Delirium | Through intervention completion, up to 4 weeks
  Proportion of participants who develop delirium, measured by the Confusion Assessment Method or the Family Confusion Assessment Method
Number of Participants With Adverse Events - Serotonin Syndrome | Through intervention completion, up to 4 weeks
  Proportion of participants who develop serotonin syndrome, diagnosed by Study Doctor
Number of Participants With Adverse Events - Adverse Mood or Behaviour Change | Measured at baseline and from enrolment to intervention completion (up to 4 weeks); 2-week and 4-week follow-up
  Proportion of participants who report adverse mood or behaviour changes (recorded daily in a participant diary)
Psychological Distress - Anxiety and Depression | Baseline
  Measured using the Hospital Anxiety and Depression Scale (higher score indicate worse anxiety/depression)
Change in Psychological Distress - Anxiety and Depression | Weekly (every Friday) during intervention (4 weeks)
  Measured using the Hospital Anxiety and Depression Scale (higher score indicate worse anxiety/depression)
Change in Psychological Distress - Anxiety and Depression | Follow-up (1 day, 2 weeks, 4 weeks, 12 weeks, 24 weeks)
  Measured using the Hospital Anxiety and Depression Scale (higher score indicate worse anxiety/depression)
Psychological Distress - Anxiety, Depression, and Well-being | Baseline
  Measured using the Edmonton Symptom Assessment System anxiety, depression, and well-being item scores (score 0-10 for each item - higher scores indicate worse symptoms)
Change in Psychological Distress - Anxiety, Depression, and Well-being | Weekly (every Friday) during intervention (4 weeks)
  Measured using the Edmonton Symptom Assessment System anxiety, depression, and well-being item scores (score 0-10 for each item - higher scores indicate worse symptoms)
Change in Psychological Distress - Anxiety, Depression, and Well-being | Follow-up (1 day, 2 weeks, 4 weeks, 12 weeks, 24 weeks)
  Measured using the Edmonton Symptom Assessment System anxiety, depression, and well-being item scores (score 0-10 for each item - higher scores indicate worse symptoms)
Psychological Distress - Global Impression of Change | Weekly (every Friday) during intervention (4 weeks); 1 day, 2 week, 4 week, 12 week, 24 week follow-up
  Measured using the Patient Global Impression of Change scale (higher scores indicate greater positive change)
Dosing | Weekly (each Friday) for intervention period (4 weeks)
  Dose at which therapeutic benefit, if any, is achieved assessed by change in Hospital Anxiety and Depression Scale score (score reduction of 50% indicates therapeutic benefit)
Dosing | Weekly (each Friday) for intervention period (4 weeks)
  Dose at which therapeutic benefit, if any, is achieved assessed by Edmonton Symptom Assessment Scale score (two-point score reduction or absolute score less than 3 indicate therapeutic benefit)
Dosing | Weekly (each Friday) for intervention period (4 weeks)
  Dose at which therapeutic benefit, if any, is achieved assessed by Global Impression fo Change score (score of 5 or above indicate therapeutic benefit)

SECONDARY OUTCOMES:
Existential Distress | Baseline (Friday prior to first dose administered on a Monday); 1 day, 2 week, 4 week, 12 week, 24 week follow-up
  Measured using the Demoralization scale II (DS-II), a 16-item questionnaire that measures loss of meaning and purpose, distress, and coping abilities. Each item is rated as a 0 (Never), 1 (Sometimes), or 2 (Often). The 16 items are then summed to create a total score. The highest total score that can be obtained is 32. Higher total scores indicate higher levels of demoralization.
Psychological distress | Baseline (Friday prior to first dose administered on a Monday); 1 day, 2 week, 4 week, 12 week, 24 week follow-up
  Measured by the Hamilton Depression Rating Scale (HDRS), a 17-item questionnaire. We will consider a 50% reduction in score from baseline as achieving clinically meaningful improvement. Each item varies in the maximum value it can be rated at (an item can be rated from 0-2, 0-3, or 0-4). The highest total score that can be obtained is 53. All scores from the 17-items are summed for a total score. Higher total scores indicate increased severity of depression.
Participant Quality of Life | Baseline (Friday prior to first dose administered on a Monday); 1 day, 2 week, 4 week, 12 week, 24 week follow-up
  Measured using the World Health Organization Quality of Life, Brief Version (higher scores indicate higher quality of life)
Wish to Die | Baseline (Friday prior to first dose administered on a Monday); 1 day, 2 week, 4 week, 12 week, 24 week follow-up
  Measured using the Categories of Attitudes Towards Death Occurrence (scored 1-6 with scores 4-6 indicating a wish to die)
Global Distress | Baseline (Friday prior to first dose administered on a Monday); 1 day, 2 week, 4 week, 12 week, 24 week follow-up
  Measured using the Distress Thermometer

CONTACTS AND LOCATIONS:
Overall Officials: James Downar, MDCM, MSc, Principal Investigator — The Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steis MR, Evans L, Hirschman KB, Hanlon A, Fick DM, Flanagan N, Inouye SK. Screening for delirium using family caregivers: convergent validity of the Family Confusion Assessment Method and interviewer-rated Confusion Assessment Method. J Am Geriatr Soc. 2012 Nov;60(11):2121-6. doi: 10.1111/j.1532-5415.2012.04200.x. Epub 2012 Oct 5. PMID 23039310
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Mitchell AJ, Meader N, Symonds P. Diagnostic validity of the Hospital Anxiety and Depression Scale (HADS) in cancer and palliative settings: a meta-analysis. J Affect Disord. 2010 Nov;126(3):335-48. doi: 10.1016/j.jad.2010.01.067. Epub 2010 Mar 5. PMID 20207007
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Watanabe SM, Nekolaichuk C, Beaumont C, Johnson L, Myers J, Strasser F. A multicenter study comparing two numerical versions of the Edmonton Symptom Assessment System in palliative care patients. J Pain Symptom Manage. 2011 Feb;41(2):456-68. doi: 10.1016/j.jpainsymman.2010.04.020. Epub 2010 Sep 15. PMID 20832987
- [Background] Galiana L, Rudilla D, Oliver A, Barreto P. The Short Demoralization Scale (SDS): A new tool to appraise demoralization in palliative care patients. Palliat Support Care. 2017 Oct;15(5):516-523. doi: 10.1017/S1478951516000973. Epub 2017 Jan 9. PMID 28065203
- [Background] Templer DI. The construction and validation of a Death Anxiety Scale. J Gen Psychol. 1970 Apr;82(2d Half):165-77. doi: 10.1080/00221309.1970.9920634. No abstract available. PMID 4394812
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] World Health Organization Division of Mental Health. WHOQOL-BREF : introduction, administration, scoring and generic version of the assessment : field trial version, December 1996. Geneva: World Health Organization; 1996
- [Background] Durst AV, Spencer B, Bula C, Fustinoni S, Mazzocato C, Rochat E, Rubli Truchard E, Monod S, Jox RJ. Wish to Die in Older Patients: Development and Validation of Two Assessment Instruments. J Am Geriatr Soc. 2020 Jun;68(6):1202-1209. doi: 10.1111/jgs.16392. Epub 2020 Feb 29. PMID 32112569
- [Background] National Comprehensive Cancer Network. NCCN Distress Thermometer and Problem List for Patients. Version 2, dated March 11th, 2020. https://www.nccn.org/about/permissions/thermometer.aspx
- [Background] Anderson F, Downing GM, Hill J, Casorso L, Lerch N. Palliative performance scale (PPS): a new tool. J Palliat Care. 1996 Spring;12(1):5-11. PMID 8857241
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Ross S, Bossis A, Guss J, Agin-Liebes G, Malone T, Cohen B, Mennenga SE, Belser A, Kalliontzi K, Babb J, Su Z, Corby P, Schmidt BL. Rapid and sustained symptom reduction following psilocybin treatment for anxiety and depression in patients with life-threatening cancer: a randomized controlled trial. J Psychopharmacol. 2016 Dec;30(12):1165-1180. doi: 10.1177/0269881116675512. PMID 27909164
- [Derived] Downar J, Lapenskie J, Anderson K, Parsons G, Polskaia N, Lalumiere G, Lawlor P. PSilocybin for psYCHological and existential distress in PALliative care (PSYCHED-PAL): A single arm unblinded clinical trial. Palliat Med. 2026 Jan 30:2692163261416269. doi: 10.1177/02692163261416269. Online ahead of print. PMID 41617652